CLINICAL TRIAL: NCT06568185
Title: The Effectiveness of Fixed Dose Combination of Alpha Lipoic Acid and Vitamin B Preparations for Treatment of Diabetic Polyneuropathy in Type 2 Diabetes Mellitus Patients: A Randomized Placebo-controlled Trial
Brief Title: The Effect of Alpha Lipoid Acid and Vitamin B Preparation on Diabetic Polyneuropathy in Type 2 Diabetes Mellitus Patient
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: BREGO Life Sciences Sdn Bhd (Unknown)
Responsible Party: Principal Investigator, Che Nur Ain binti Che Abdullah, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23110893
Record Dates: First submitted 2024-05-06; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Intervention Model Description: The participants then will be randomized to either intervention or control group. The intervention group will receive a fixed dose combination of alpha lipoic acid and vitamin B preparations, and the control group will receive a placebo (look-alike substance that contains no drug).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bionerve (Experimental): The participants will receive a fixed dose combination of alpha lipoic acid and vitamin B preparations.
  Interventions: Drug: Alpha-Lipoic Acid/Vitamin/Mineral Supplement PolyMVA
- Placebo (No Intervention): The participants will receive a placebo (look-alike substance that contains no drug)l

INTERVENTIONS:
Drug: Alpha-Lipoic Acid/Vitamin/Mineral Supplement PolyMVA — BIONERV® s the first combination of alpha lipoic acid 300mg and vitamin B complex. Bionerv® is in oral film-coated, orange colour, oblong shape and no marking and embossing on the tablet. Each tablet contains 4 active ingredients as follows: Alpha lipoic acid 300mg, Vitamin B12 (methylcobalamin) 500mcg, Vitamin B6 (pyridoxine) 8mg, Vitamin B1 (thiamine) 39mg. To be taken after meal 1 tablet once daily.
  Other Names: BIONERV
  Arms: Bionerve

SUMMARY:
To evaluate the efficacy of combination of vitamin B and alpha lipoic acid formulations for the treatment of diabetic polyneuropathy in individuals with type 2 diabetes mellitus.

Methodology :

This is a single-center, randomized, double-blind, placebo-controlled trial study.

Study duration May 2024 - September 2025

Study location :

This study will be conducted at the Klinik Rawatan Keluarga and diabetes clinic Hospital Universiti Sains Malaysia.

Source Reference :

People with type 2 diabetes mellitus attending the Hospital Universiti Sains Malaysia.

Study source population :

People with type 2 diabetes mellitus attended Klinik Rawatan Keluarga and diabetes clinic Hospital Universiti Sains Malaysia during the study period.

DETAILED DESCRIPTION:
General objective

To determine the effectiveness of a fixed dose combination of alpha lipoic acid and vitamin B preparations in comparison with incative drug for treatment of diabetic polyneuropathy (DPN) in people with type 2 diabetes mellitus.

Research hypothesis

1. There are significant improvements in mean total symptom score (TSS) and neuropathic symptoms score (NSS) in people with diabetic polyneuropathy taking a fixed dose combination of alpha lipoic acid and vitamin B preparations as compared to diabetic polyneuropathy patients taking a placebo.
2. There are significant improvements in total symptom score (TSS) and neuropathic symptoms score (NSS) among people with diabetic polyneuropathy taking a fixed dose combination of alpha lipoic acid and vitamin B preparations for 12 weeks.
3. There are significant improvements in fasting plasma glucose, HbA1C level, fasting lipid profile, body mass index (BMI), and diabetes quality of life in people with diabetes taking a fixed dose combination of alpha lipoic acid and vitamin B preparations as compared to diabetic patients taking placebo.
4. There are no significant differences in the safety parameters of renal function and liver function tests among people with diabetic polyneuropathy at baseline and 12 weeks after taking a fixed dose combination of alpha lipoic acid and vitamin B preparations.
5. There are significant improvements in fasting plasma glucose, HbA1C level, fasting lipid profile, body mass index (BMI), and diabetes quality of life among diabetic patients taking a fixed dose combination of alpha lipoic acid and vitamin B preparations for 12 weeks.

Method of data collection

This study will be conducted after obtaining approval from the Universiti Sains Malaysia Ethical Committee (JPeM) and will be conducted in accordance to World Medical Association Declaration of Helsinki ethical principles for medical research involving human subjects.

Recruitment of subject

Participants will be recruited from Klinik Rawatan Keluarga and diabetes clinic Hospital USM via convenience sampling. Potential participants will be identified from the case notes of patients. Then, the participants will be approached individually. Those who are willing to participate in this study will be given information regarding the study. The participants will be screened to determine their eligibility criteria, including performing neurological symptom score (NSS) and neuropathy disability score (NDS) to determine diabetes polyneuropathy diagnosis. If all the inclusion and exclusion criteria are fulfilled, informed consent will be obtained from all patients who agree to participate in this study. The consent will be obtained by a study team that recruited the patient. Upon consented, the participant's socio-demographic data will be collected, and the medical record will be assessed to fill in their medical and diabetes profiles. They will also answer the total symptoms score (TSS), and revised version of the Diabetes Quality of Life (Rv-DQoL) questionnaire. The physical examination includes measurement of height, weight, calculated Body Mass Index (BMI), and blood pressure during sitting will be done. Then 6ml of fasting venous blood will be taken for measurement of HbA1c, fasting blood glucose, renal function test, liver function test and fasting lipid profile as baseline. All participants were advised not to consume any special supplement or other replacement meal throughout the study.

The participants then will be randomized to either intervention or control group. The intervention group will receive a fixed dose combination of alpha lipoic acid and vitamin B preparations, and the control group will receive a placebo (look-alike substance that contains no drug).

The participants will be seen 6 weeks after taking the product. During this visit, they will be assessed for any side effects or adverse events and compliance with the product supplied (compliance form). The total symptoms score (TSS), neurological symptom score (NSS), a revised version of Diabetes Quality of Life (Rv-DQoL), blood pressure, weight, height, calculated Body Mass Index (BMI) will also be measured. Another 6-week supply of the product will be given.

Lastly, the participants will be assessed in week 12. During this visit, the same measurement will be taken as visit 1, including answering the questionnaires. Adverse events, blood taking, and compliance will also be assessed.

The duration for visit 1 and visit 3 (at 12 weeks) is about 50-60 minutes for each visit since it will involve blood taking procedure. Duration for visit 2 (at 6 weeks) is about 30 minutes since it will not involve blood taking.

Intervention group: Fixed dose combination of alpha lipoic acid and vitamin B preparations

At baseline, the intervention group will receive a fixed dose combination of alpha lipoic acid and vitamin B preparations. This product is packaged and manufactured by BREGO Life Sciences Sdn Bhd company with a brand name of Bionerv®. BIONERV® is the first combination of alpha lipoic acid 300mg and vitamin B complex. Bionerv® is in oral film-coated, orange colour, oblong shape and no marking and embossing on the tablet. Each tablet contains 4 active ingredients as follows: Alpha lipoic acid 300mg, Vitamin B12 (methylcobalamin) 500mcg, Vitamin B6 (pyridoxine) 8mg, Vitamin B1 (thiamine) 39mg. All the above ingredients are synthetic. The shelf-life is 2 years. Storage condition is keeping in dry place below 300oC and protecting from light and moisture. It has no bovine-gelatin capsule. There are no precautions on drug-drug interaction, but it is not suitable for children (<18 years). There is insufficient reliable data for pregnancy and breast feeding. One bottle consists of 60 tablets.

This medication needs to take 2 tablets a day after a meal and need to drink more water. In this study, the participants need to take 2 tablets once daily after breakfast. The duration of the intervention will be 12 weeks. All participants are required to return to the clinic in the 6th and 12th week for a post-intervention assessment.

Control group

At baseline, the control group will receive a placebo drug consisting of Croscamellose Sodium, Microcrystalline Cellulose, Silicon Dioxide and Magnesium stearate. The placebo was manufactured by Yanling Natural Hygiene Sdn Bhd. The formulation of the placebo tablet is derived from the excipients used in the Bionerv tablet.

The participants need to take 2 tablets once daily after breakfast. The placebo drugs will share the same appearance and color as intervention drug.

The duration of the intervention will be 12 weeks. All participants are required to return to the clinic in the 6th and 12th week for a post-intervention assessment.

Follow up

There are two follow-ups during this study. 1st follow-up will be on the 6th week and 2nd follow-up (final follow-up) will be during 12th week of the study.

During the 6th week follow-up, participants will be checked for their weight, height, calculated Body Mass Index (BMI), TSS, NSS, RV-DQoL questionnaire, compliance, and adverse effects.

A final visit (12th week) to the clinic will be conducted on the 12th week. During these visits, the outcome measures will be assessed to determine the effect of the fixed-dose combination of alpha lipoic acid and vitamin B. During this visit, the same measurement will be taken as visit 1.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and over
2. Diagnosed with type 2 diabetes mellitus based on WHO diagnostic criteria for diabetes (Organization, 2020).
3. Diagnose with diabetic polyneuropathy by Neurological Symptom Score (NSS) and Neuropathy Disability Score (NDS).

Exclusion Criteria:

1. Those with a documented mental impairment which impacted on their ability to answer questions independently.
2. People with peripheral vascular disease (non-palpable foot pulses, intermittent claudication)
3. People with an amputated foot or leg
4. Abnormal liver enzyme.
5. People with renal impairment.
6. People using drugs with possible influence on the study results (antidepressants, anticonvulsants, opiates, neuroleptics, antioxidants, and particularly methylcobalamin, pyridoxine and other B complex preparations)
7. Pregnancy, lactation, or childbearing age without safe contraception
8. History of allergy with vitamin B complex preparations (i.e. Vitamin B12, B6 and B1) and alpha lipoic acid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
To compare the mean change in Total symptom score (TSS) over 12 a week period | baseline, 6 weeks and 3 month
  Total Symptom Score is the sum of 4 neuropathic symptoms (stabbing pain, burning pain, paraesthesia, and numbness) reported as symptoms frequency (occasionally, frequent, or continuous) and symptom intensity (absent, slight, moderate, or severe) on which scores range from 0 to 14.64.
To compare the mean change in Neuropathic symptoms score (NSS) over 12 a week period | baseline, 6 weeks and 3 month
  Neurological Symptom Score consists of 4 components. The first component is on reported discomfort symptoms: burning/numbness/tingling (2 points), fatigue/cramping and aching feelings (1point) and 0 point for none. Second component is on symptom location whether the symptom occurs in the feet (2 points), calves (1 point) and 0 points for elsewhere. The third component is on timing of symptoms, either nocturnal exacerbation (2 points), symptoms present both day and night (1 point) and 0 for symptoms present during daytime only. A score of 1 was added if the symptoms had ever woken the patient from sleep. The fourth component is on a manoeuvre to reduce the symptoms by either walking (2 points) or standing (1pointand and 0 for sitting or lying down. The maximum symptom score was 9.

SECONDARY OUTCOMES:
compare the changes in the fasting plasma glucose over 12 a week period | baseline and 3 month
  A fasting blood glucose test measures the amount of glucose in blood after a period of fasting (usually 8-12 hours). Fasting plasma glucose will be measure in millimoles per liter (mmol/L). The participants fasts overnight, usually for 8 hours before the test.
compare the changes in the fasting lipid profile over 12 a week period | baseline and 3 month
  A fasting lipid profile (or lipid panel) measures the levels of various types of fats in the blood, including Total Cholesterol, High-Density Lipoprotein (HDL) Cholesterol, Low-Density Lipoprotein (LDL) Cholesterol and triglycerides. Fasting lipid profile will be measure in millimoles per liter (mmol/L). Patients are usually advised to fast overnight, avoiding food and drinks (except water) for 8 hours before the test.
compare the changes in the HbAIC level over 12 a week period | baseline and 3 month
  The HbA1c test reflects the average blood glucose levels by measuring the percentage of glycated hemoglobin (hemoglobin bound with glucose) and is an important indicator of long-term blood sugar control. The HbA1c results are reported as a percentage (%) of glycated hemoglobin. The target HbA1C level for most diabetic individuals is typically below 7% to reduce the risk of diabetes-related complications.
compare the changes in blood pressure over 12 a week period | baseline and 3 month
  A blood pressure cuff is placed around the upper arm and inflated. The cuff then deflates while measuring the pressure in the arteries. The measurement is taken with an electronic sphygmomanometer. Blood pressure is measured in millimeters of mercury (mmHg). Normal Blood Pressure is systolic less than 120 mmHg and diastolic less than 80 mmHg.
compare the changes in diabetes quality of life over 12 a week period | baseline, 6 weeks and 3 month
  using the revised version of Diabetes Quality of Life (Rv-DQoL) questionnaire. DQoL used for evaluating the quality of life specifically related to Type 2 Diabetes Mellitus patient and was made up of three major domains, namely, (i) Diabetes Life Satisfaction (QoL Satisfy), 18 items; (ii) Disease Impact Scale (QoL Impact), 27 items; and (iii) Disease-Related Worries Scale (QoL Worry), 14 items and one general question to reflect self-rating of overall general health. All items in the QoL Satisfy domain are scored on a five-point scale, ranging from 1 (very satisfied) to 5 (very dissatisfied), whereas the items in the QoL Impact and QoL Worry are scored on a five-point scale, ranging from 1 (never) to 5 (all the time); the score was presented as the total of the items of each scale divided by the number of items. A higher average score indicates poorer QoL.
compare the differences in the safety parameters of renal function | baseline and 3 month
  The test conducted to assess kidney function include Blood Urea Nitrogen (BUN), Serum Creatinine and Estimated Glomerular Filtration Rate (eGFR). Blood Urea Nitrogen (BUN) measure in mg/dL which the Normal Range: 7 to 20 mg/dL. Serum Creatinine measure in Micromoles per liter (µmol/L) Normal Range for Men: Approximately 70 to 120 µmol/L while Women: Approximately 50 to 100 µmol/L. Estimated Glomerular Filtration Rate (eGFR) normal range: 90 to 120 mL/min/1.73 m². Values below 60 mL/min/1.73 m² suggest CKD (Chronic Kidney Disease).
compare the differences in the safety parameters of liver function | baseline and 3 month
  Liver function tests (LFTs) in encompass a range of blood tests that assess the health and function of the liver. This include: 1) Alanine Aminotransferase (ALT) which typically below 40 international units per liter (IU/L) for men and below 30 IU/L for women. 2) Aspartate Aminotransferase (AST) with normal range usually below 40 IU/L for both men and women. 3) Alkaline Phosphatase (ALP) varies by age and gender, typically between 30 and 120 IU/L.
compare the changes in participant weight. | baseline, 6 weeks and 3 month
  participant weight will be measure in kilograms (kg) using electronic bathroom scale.
participant height. | baseline
  participant height measurement will be measure using a stadiometer. It consists of a vertical ruler and a movable headpiece that is adjusted to rest on the top of the head. Height measurement is in Centimeters (cm).
compare the changes in participant Body Mass Index (BMI) | baseline, 6 weeks and 3 month
  Body Mass Index (BMI) is used to measure whether a person is underweight, normal weight, overweight, or obese. It is calculated by dividing weight in kilograms by height in meters squared (BMI = weight(kg) / height(m)^2). In Malaysia, the Clinical Practice Guidelines (CPG) on the Management of Obesity provide specific classifications for Body Mass Index (BMI) to identify and manage obesity. Underweight: BMI < 18.5. Normal Weight: BMI 18.5-22.9. Overweight: BMI 23.0-27.4. Obesity Class I: BMI 27.5-34.9. Obesity Class II: BMI 35.0-39.9. Obesity Class III (Morbid Obesity): BMI ≥ 40.0.

CONTACTS AND LOCATIONS:
Overall Officials: Che Nur Ain Che Abdullah, Dr., Principal Investigator — Department of Family Medicine, School of Medical Sciences University Sains Malaysia, Health Campus; Noraini Mohamad, Dr., Study Director — Department of Family Medicine, School of Medical Sciences University Sains Malaysia, Health Campus; Nani Draman, Prof. Dr., Study Chair — Department of Family Medicine, School of Medical Sciences University Sains Malaysia, Health Campus; Ritzzaleena Rosli Mohd Rosli, Dr., Study Chair — Department of Family Medicine, School of Medical Sciences University Sains Malaysia, Health Campus; Zainab Mat Yudin@Badrin, Dr., Study Chair — Department of Family Medicine, School of Medical Sciences University Sains Malaysia, Health Campus
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT06568185/Prot_SAP_000.pdf
  • Informed Consent Form: INFORMED CONSENT BIONERV STUDY (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT06568185/ICF_001.pdf
  • Informed Consent Form: CRF BIONERV STUDY (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT06568185/ICF_002.pdf